CLINICAL TRIAL: NCT00003360
Title: Phase I Study of 131I-Labeled Humanized Antibody A33 in Patients With Advanced Colorectal Carcinoma
Brief Title: Radiolabeled Monoclonal Antibody in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-011; MSKCC-98011; NCI-H98-0017
Record Dates: First submitted 1999-11-01; First posted 2004-08-16 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody A33

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and deliver tumor-killing substances, such as radioactive iodine, to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody in treating patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the toxicity and determine the maximum tolerated dose of iodine I 131 humanized monoclonal antibody A33 (131I-huAb A33) in patients with advanced colorectal cancer. II. Describe pharmacokinetics and biodistribution of 131I-huAb A33 by external imaging in these patients. III. Determine the effect of human antihuman antibody response on pharmacokinetics and targeting of 131I-huAb A33 in this patient population. IV. Determine whether the dose planning methodology used here can adequately and safely be applied to routine radioimmunotherapy planning.

OUTLINE: Patients receive iodine I 131 humanized monoclonal antibody A33 (131I-huAb A33) by IV infusion over 20 minutes every 6-8 days for up to 8 weeks (depending on dosage). Patients receive a minimum of 6 weeks of treatments. In the absence of disease progression or unacceptable toxicity, patients are retreated no sooner than 6 weeks after the previous course. Cohorts of 3-6 patients receive escalating doses of 131I-huAb A33 to determine the maximum tolerated dose (MTD). The MTD is defined as the highest dose at which no more than 2 of 6 patients experience dose limiting toxicity. Patients are followed for 6 weeks after the last treatment.

PROJECTED ACCRUAL: There will be 3-24 patients accrued into this study over 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced colorectal cancer Must have unresectable (Stage IV) disease or have failed or refused conventional chemotherapy Measurable disease by conventional imaging methods Liver involvement no greater than 50% No CNS involvement Not positive for human antimouse antibody titer

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 80-100% Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 150,000/mm3 Prothrombin time less than 1.3 times control Hepatic: Bilirubin no greater than 1 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No significant cardiac disease (New York Heart Association class II/IV heart disease) Other: No serious infection requiring treatment with antibiotics No other serious illness Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior mouse monoclonal antibody or antibody fragment, chimeric or humanized antibody, or constructs derived from antibodies At least 4 weeks since prior immunotherapy Chemotherapy: No prior mitomycin/radiotherapy combination At least 4 weeks since prior chemotherapy Endocrine therapy: No concurrent steroids or other antiinflammatory agents Radiotherapy: No prior radiotherapy/mitomycin combination Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1998-04; Primary Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Welt, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States